CLINICAL TRIAL: NCT06064604
Title: Clinical Trial: Powered Hip & Ankle Exoskeletons for Stroke Survivors With Gait Impairment
Brief Title: Clinical Efficacy of Exoskeleton Assistance for Individuals Post-Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H23332; R01HD113598-01 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stoke; Robotic Exoskeleton; Gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study includes one pre-specified group, stroke survivors, to receive intervention with two exoskeleton devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stroke Survivors (Experimental): This study will be divided into 2 sessions that will occur on 2 separate days: 1) Hip Exoskeleton session and 2) Ankle Exoskeleton session. In each session, subjects will undergo two conditions in which they complete the outcomes measures 1) while wearing the exoskeleton and 2) in a baseline condition without the exoskeleton. Order of condition and session will be randomized.
  Prior to the exoskeleton condition, subjects will be allowed time to acclimate to the device during a walking session on the treadmill. Subjects will complete several timed walking tests both indoors and outdoors. Measurements of energy expenditure may also be recorded along with patient reported outcomes data to assess participant perception of their performance with and without the devices.
  Interventions: Other: Control; Device: Hip Exoskeleton; Device: Ankle Exoskeleton

INTERVENTIONS:
Other: Control — The stroke survivors will serve as their own control group. The participants will complete the required tasks without an exoskeleton device.
  Other Names: No-exoskeleton
Device: Hip Exoskeleton — The Georgia Tech Hip Exo is a wearable robotic device for hip extension/flexion assistance. This device will be used to study the lower limb movement and how to effectively assist users. It makes use of a responsive controller that considers information such as joint angles to understand the user's state and assists with the appropriate level of power accordingly.
  Other Names: Georgia Tech Hip Expo
Device: Ankle Exoskeleton — The Dephy Exoboot is a lower limb exoskeleton which attaches to the user below the knee through a cuff at the proximal calf and a provided shoe. This investigational device is used to make it easier for able-bodied and impaired individuals to walk and run under a variety of conditions. The exoskeleton provides assistance at the ankle joint during movement. The purpose is to assist the user in lower limb movements such as ground level walking, climbing stairs/ramps, and sit-to-stand.
  Other Names: Dephy ExoBoot

SUMMARY:
An exoskeleton device is a robotic system designed to improve an individual's ability to move and perform tasks encountered in everyday situations. These devices consist of external rigid limb segments that assists humans through different body movements with the use of actuators. These devices are controlled by an onboard computer that determines the timing and magnitude of assistance deployed to the user. Exoskeleton controller performance is key to providing beneficial assistance that does not inhibit the user's movement. Preceding work will compare the benefit of personalized hip versus ankle joint exoskeleton assistance for improvement of post-stroke gait. It will combine exoskeleton technology with the user's movement feedback to improve wearable robotic assistance to an individual stroke survivor's gait pattern. For the clinical trial research covered under this protocol, the investigator will test various exoskeleton technologies with stroke survivors in real-world contexts, indoors and outdoors, and measure clinically meaningful outcomes and user perceptions regarding technology usability and adoption. The long-term goal is to deploy self-adaptive, adoptable exoskeletons for personalized assistance during community ambulation.

DETAILED DESCRIPTION:
Participants will serve as their own control in this study. This study will be divided into 2 sessions that will occur on 2 separate days: 1) Hip Exoskeleton session and 2) Ankle Exoskeleton session. In each session, subjects will undergo two conditions in which they complete the outcomes measures 1) while wearing the exoskeleton and 2) in a baseline condition without the exoskeleton. Order of condition and session will be randomized.

Prior to the exoskeleton condition, subjects will be allowed time to acclimate to the device during a walking session on the treadmill. Subjects will proceed to complete a timed indoor community circuit in which they will complete a 10 meter walk test over an instrumented gait mat which will record information about their walking. The indoor community circuit may also include turning, walking up/down a ramp and walking up/down a staircase.

Subjects will then proceed to complete an outdoor 6-minute walk test (6MWT) on a pre-defined course on Georgia Tech's campus. When outdoors, participants will be guarded with a gait belt and a researcher who will walk alongside them throughout the experiment to reduce the risk for a fall. Borg Rating of Perceived Exertion (RPE) and Physiological Cost Index (PCI) will be assessed and calculated following completion of the 6MWT. Following each condition, subjects will then sit, rest and complete a suite of patient reported outcomes in which the investigators will ask questions about their perception of their performance with and without the device; investigators will also ask them questions about the device. Following completion of surveys, subjects will repeat the same outcomes for the other condition- either the baseline condition or the exoskeleton condition, depending on the initial randomization.

Throughout the procedures, subjects will be monitored for fatigue and asked if they need a break. They will be encouraged to voice any concerns (discomfort, fatigue or otherwise) to the research personnel, who will respond accordingly. Participants will be guarded with a gait belt or harness to reduce the risk of falls while participating in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-85 years of age
* Stroke at least 6 months prior to study involvement
* Community dwelling (participant does not live in an assisted living facility)
* Able to provide informed consent to participate in the study activities
* Can safely participate in the study activities (per self-report)
* Must have a Functional Ambulation Category (FAC) score of 3 or above (the participant can walk without the assistance of another person)

Exclusion Criteria:

* Requires a walker to walk independently
* Has a shuffling gait pattern overground
* Has a Functional Ambulation Category (FAC) score of 2 or lower (the participant requires the assistance of another person in order to walk)
* Has a significant secondary deficit beyond stroke (e.g. amputation, legal blindness or other severe impairment or condition) that in the opinion of the Principal Investigator (PI), would likely affect the study outcome or confound the results
* For exoskeleton-only studies, the exoskeleton device does not fit appropriately or safely, as determined by the research team during the fitting assessment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test (10MWT) | 2 weeks
  This measures the individual's preferred overground walking speed, indicating their physical capability with an exoskeleton device
6-minute walk test (6MWT) | 2 weeks
  This measures the individual's walking distance over 6 minutes to assess aerobic endurance.
Physiological Cost Index | 2 weeks
  This measures the individual's oxygen consumption while walking. It will be calculated using a 6-minute walk test (6MWT) and heart rate.
Borg Rating of Perceived Exertion (RPE) | 2 weeks
  This measures the individual's perceived physical activity intensity level, indicating how hard the individuals believes their body is working to conduct walking tasks with and without the exoskeleton devices.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Young, PhD, Principal Investigator — Georgia Institute of Technology; Greg Sawicki, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Exoskeleton and Prosthetic Intelligent Controls Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No